CLINICAL TRIAL: NCT01406119
Title: An Extension Study of ABT-806 for Subjects With Advanced Solid Tumors
Brief Title: An Extension Study of ABT-806 in Subjects With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AbbVie (prior sponsor, Abbott) (Industry)
Responsible Party: Sponsor
Organization: AbbVie (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M12-326
Record Dates: First submitted 2011-07-28; First posted 2011-08-01 (Estimated); Last update posted 2017-01-27 (Estimated); Status verified 2017-01

CONDITIONS: Advanced Solid Tumors
MeSH Terms: interventions — depatuxizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ABT-806 Arm (Experimental)
  Interventions: Drug: ABT-806

INTERVENTIONS:
Drug: ABT-806 — ABT-806 will be administered by intravenous infusion.

SUMMARY:
This is an extension study of ABT-806 for subjects with advanced solid tumors.

ELIGIBILITY:
Inclusion Criteria:

* Subject has completed a prior study utilizing ABT-806 or 111ln ABT-806 (ABT 806i) and the Investigator believes that continued treatment with ABT-806 is in the best interest of the subject.
* Women of childbearing potential and men must agree to use adequate contraception (one of the following listed below) prior to study entry, for the duration of study participation and for a period of 3 months. Female subjects considered not of childbearing potential must be documented as being surgically sterile or post-menopausal for at least 1 year.
* Subject is capable of understanding and complying with parameters as outlined in the protocol and the subject or the subject's legal acceptable representative is able to sign informed consent, approved by an Institutional Review Board (IRB) prior to the initiation of any or study-specific procedures.

Exclusion Criteria:

* Subject discontinued ABT-806 or111ln ABT-806 (ABT-806i) administration before completing the prior study (due to disease progression, toxicity, withdrawn consent, other).
* Subject has any medical condition which in the opinion of the investigator places the subject at an unacceptably high risk for toxicities.
* Subject is a lactating or pregnant female.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2011-10; Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Safety (Number of subjects with adverse events) | At each treatment visit (every other week throughout the study or up to 51 weeks)
  Evaluation of vitals signs, clinical lab testing and adverse event monitoring (every other week), physical exam (every 4 weeks) and ECG (at final visit)
Pharmacokinetic profile (assay for ABT-806) | Every 8 weeks starting at Week 9 throughout the study or up to 51 weeks
  Assay for ABT-806

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Ocampo, MD, Study Director — AbbVie
Locations (4):
- United States (2):
  - Site Reference ID/Investigator# 58883, Baltimore, Maryland
  - Site Reference ID/Investigator# 58882, Boston, Massachusetts
- Australia (2):
  - Site Reference ID/Investigator# 60619, Heidelberg
  - Site Reference ID/Investigator# 63845, Herston